CLINICAL TRIAL: NCT06625242
Title: A Multicenter, Open-label, Single-arm, Phase 4 Study to Evaluate the Efficacy and Safety of Filgotinib in Korean Patients With Rheumatoid Arthritis
Brief Title: A Study of Filgotinib in Korean Participants With Rheumatoid Arthritis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS6034-M082-401
Record Dates: First submitted 2024-09-30; First posted 2024-10-03 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Filgotinib Maleate
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Filgotinib Maleate 100 or 200 milligram (Experimental)
  Interventions: Drug: Filgotinib Maleate

INTERVENTIONS:
Drug: Filgotinib Maleate — Administered as oral tablets.
  Other Names: Jyseleca

SUMMARY:
The primary purpose of this study is to assess the percentage of participants achieving an American College of Rheumatology (ACR) 20 percent (%) Improvement (ACR20) response at Week 12 of the administration of the investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who voluntarily provided written consent to participate in this study
2. Male or female, aged greater than or equal to (>=) 19 years at the time of written informed consent
3. Participants diagnosed with rheumatoid arthritis according to the 2010 ACR/ European League Against Rheumatism (EULAR) classification criteria and who have an ACR functional class of I to III
4. Participants who meet the following criteria are eligible for the specified treatment protocol; those who have been treated with two or more type types (including MTX) of Disease-Modifying Antirheumatic Drugs (DMARDs) for at least 6 months (at least 3 months each) but have experienced insufficient therapeutic effects or have had to discontinue treatment due to adverse events of these medications (However, in cases where MTX is contraindicated due to conditions such as liver disease or renal failure, the participant must have been treated with at least two types of DMARDs, excluding MTX).

   * Furthermore, in participants over 65 years of age, those at high risk of cardiovascular diseases, and those with a potential risk of malignancy, this protocol applies if they have not adequately responded to or tolerated conventional therapies, including Tumor Necrosis Factor (TNF) inhibitors or other biologic agents. Eligibility is confirmed if one of the following criteria is met:

     1. DAS28 score exceeding 5.1.
     2. DAS28 score between 3.2 and 5.1, with diagnostic imaging showing progression of joint damage.

Exclusion Criteria:

1. Participants with hypersensitivity reactions to the active ingredient or other components of the investigational product
2. Participants with serious infections (for example [e.g.], sepsis) or active infections including localized infections
3. Participants with active tuberculosis (TB)
4. Participants with severe hepatic impairment (e.g., Child-Pugh C)
5. Participants with end-stage renal disease (<creatinine clearance [CrCl] 15 milliliters per minute [mL/min])
6. Participants with absolute neutrophil count (ANC) <1*10^9 cells per liter (/L)
7. Participants with absolute lymphocyte count (ALC) <0.5*10^9 cells/L
8. Participants with hemoglobin <8 grams per deciliter (g/dL)
9. Pregnant or lactating women
10. Women of childbearing potential who are not willing to consent to using effective contraception
11. Participants with rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption should not take this medicinal product
12. Participants who received Janus kinase (JAK) inhibitors for the treatment of rheumatoid arthritis
13. Participants who have participated in other clinical studies for investigational product/medical device within 4 weeks prior to screening
14. Participants in whom the administration of Jyseleca Tablet is contraindicated according to the product label approved in Korea or based on certain medical conditions that have been identified in previous clinical studies
15. Participants for whom follow-up deems impossible

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving ACR20 Response at Week 12 | At Week 12

SECONDARY OUTCOMES:
Percentage of Participants Achieving Disease Activity Score for 28 (DAS28) C-reactive Protein (CRP) Less Than or Equal to (<=) 3.2 at Weeks 12 and 24 | At Weeks 12 and 24
Change From Baseline in DAS28 (CRP) at Weeks 12 and 24 | Baseline, Weeks 12 and 24
Percentage of Participants Achieving DAS28 (CRP) Less Than (<) 2.6 at Weeks 12 and 24 | At Weeks 12 and 24
Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Weeks 12 and 24 | Baseline, Weeks 12 and 24
Percentage of Participants Achieving an ACR20 Response at Week 24 | At Week 24
Percentage of Participants Achieving an ACR50 and ACR70 Responses at Weeks 12 and 24 | At Weeks 12 and 24
Percentage of Participants Achieving an ACR20, ACR50 and ACR70 Responses at Week 12 and Week 24 Depending on the Prior Treatment Therapy | At Weeks 12 and 24
Percentage of Participants Achieving an ACR20, ACR50 and ACR70 Responses at Weeks 12 and 24 Depending on Monotherapy With the Investigational Product and Combination Therapy With Methotrexate (MTX) | At Weeks 12 and 24
Percentage of Participants Achieving an ACR20 Response at Week 12 Depending on Demographic Characteristics | At Weeks 12
Number of Participants With Adverse Events (AEs) | Baseline up to 28 weeks

CONTACTS AND LOCATIONS:
Locations (15):
- South Korea (15):
  - Eisai site #11, Anyang-si
  - Eisai site #01, Busan
  - Eisai site #09, Daegu
  - Eisai site #12, Daegu
  - Eisai site #06, Daejeon
  - Eisai site #15, Guri-si
  - Eisai site #02, Gwangju
  - Eisai site #13, Incheon
  - Eisai site #03, Seoul
  - Eisai site #04, Seoul
  - Eisai site #05, Seoul
  - Eisai site #07, Seoul
  - Eisai site #08, Seoul
  - Eisai site #10, Seoul
  - Eisai site #14, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.